CLINICAL TRIAL: NCT00380185
Title: The Genetic Determinants of Peripheral Arterial Disease
Brief Title: Understanding the Genetic Basis of Atherosclerosis and Peripheral Arterial Disease
Acronym: GenePAD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John P Cooke, MD, Professor of Medicine, Stanford University
Other Study IDs: 1361; R01HL075774 (NIH)
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral Arterial Disease; Atherosclerosis
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, White Cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Subjects with no hemodynamically significant disease (NHSD) of the coronary or peripheral arteries
- 2: Subjects with coronary artery disease only
- 3: Subjects with both coronary artery disease and peripheral arterial disease

SUMMARY:
Atherosclerosis, a condition in which fatty deposits build up along the inner walls of arteries, can occur throughout the body. The purpose of this study is to examine the possible genetic differences that may influence where atherosclerosis occurs.

DETAILED DESCRIPTION:
Plaque build-up caused by atherosclerosis increases the risk of blood clots, heart attack, and stroke. Blockages of plaque can occur in different areas of the body. PAD, a circulatory disorder in which blockages occur in the peripheral arteries, is one manifestation of atherosclerosis. Individuals with PAD experience reduced blood flow to the legs, which may cause leg pain while walking. Coronary artery disease (CAD), in which plaque builds up in arteries leading to the heart, is another atherosclerosis-related condition. Individuals with PAD and CAD have similar atherosclerosis risk factors, but it remains unknown why some individuals develop one disease and not the other. Genetic differences may influence where atherosclerosis develops. The goal of the study is to identify genetic variations that may cause inherited differences in plaque distribution.

This study will enroll individuals with PAD who have been referred by their doctor for a coronary angiogram to confirm the presence of CAD. A control group composed of individuals who do not have PAD, but have similar risk factors for atherosclerosis, will also be enrolled. All participants will attend one study visit. They will undergo a coronary angiogram, a procedure in which a special dye is inserted intravenously into an artery of the heart. X-rays will be taken to document how blood flows through the artery. Questionnaires assessing quality of life, exercise habits, tobacco exposure, and family medical history will be completed. Participants will also undergo blood pressure measurements and blood collection for genetic analysis. Yearly follow-up phone calls will occur for 5 years to document any hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically significant PAD, as documented by an ankle-brachial index less than 0.9; control group participants will not have PAD
* Received a referral for an elective coronary angiogram
* Suspected CAD

Exclusion Criteria:

* History of radiation treatment
* History of organ transplant
* History of viral diseases (i.e. HIV, hepatitis)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from individuals undergoing elective coronary angiography for suspected CAD at Stanford University or Mount Sinai Medical Centers.
Sampling Method: Non-Probability Sample
Enrollment: 1789 (Actual)
Dates: Start 2004-04; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Identifying genetic variations that may cause inherited differences in plaque distribution | Measured at participants' study visit

CONTACTS AND LOCATIONS:
Overall Officials: John P. Cooke, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Mt. Sinai Medical Center, New York, New York

REFERENCES:
- [Derived] Flores AM, Schuler A, Eberhard AV, Olin JW, Cooke JP, Leeper NJ, Shah NH, Ross EG. Unsupervised Learning for Automated Detection of Coronary Artery Disease Subgroups. J Am Heart Assoc. 2021 Dec 7;10(23):e021976. doi: 10.1161/JAHA.121.021976. Epub 2021 Nov 30. PMID 34845917
- [Derived] Sadrzadeh Rafie AH, Stefanick ML, Sims ST, Phan T, Higgins M, Gabriel A, Assimes T, Narasimhan B, Nead KT, Myers J, Olin J, Cooke JP. Sex differences in the prevalence of peripheral artery disease in patients undergoing coronary catheterization. Vasc Med. 2010 Dec;15(6):443-50. doi: 10.1177/1358863X10388345. PMID 21183651